CLINICAL TRIAL: NCT06864013
Title: Short-course Neoadjuvant Radiotherapy Combined With Chemotherapy and Iparomlimab and Tuvonralimab in Microsatellite Stability (MSS) or Mismatch-repair-proficient (pMMR) Patients With Locally Advanced Rectal Cancer: A Randomized Controlled Clinical Study
Brief Title: SCRT Combined With Chemotherapy and Iparomlimab and Tuvonralimab in MSS or pMMR Patients With Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ningbo No.2 Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Second Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other); The Affiliated People's Hospital of Ningbo University (Other Government); Taizhou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240172C
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Rectal Cancer (LARC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): The experimental group will receive neoadjuvant short-course radiotherapy, followed by CAPEOX+Iparomlimab and Tuvonralimab for 4 cycles. Patients who undergo surgery will receive CAPEOX combined with Iparomlimab and Tuvonralimab for 4 cycles, followed by sequential treatment with Iparomlimab and Tuvonralimab for up to 1 year.
  Interventions: Drug: Experimental
- Control Arm (Other): The control group will receive neoadjuvant short-course radiotherapy,followed by CAPEOX for 4 cycles. Patients who undergo sugery will receive CAPEOX for 4 cycles.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Experimental — The experimental group will receive neoadjuvant short-course radiotherapy (dose 25Gy/5f), followed by CAPEOX+Iparomlimab and Tuvonralimab (capecitabine 1000mg/m2 bid po d1-d14, q3w; oxaliplatin 130mg/m2 iv d1, q3w; Iparomlimab and Tuvonralimab 5mg/kg iv d1, q3w) for 4 cycles. Patients who undergo surgery will receive CAPEOX combined with Iparomlimab and Tuvonralimab for 4 cycles, followed by sequential treatment with Iparomlimab and Tuvonralimab for up to 1 year.
  Arms: Experimental Arm
Drug: Control — The control group will receive neoadjuvant short-course radiotherapy,followed by CAPEOX (capecitabine 1000mg/m2 bid po d1-d14, q3w; oxaliplatin 130mg/m2 iv d1, q3w) for 4 cycles. Patients who undergo sugery will receive CAPEOX for 4 cycles.
  Arms: Control Arm

SUMMARY:
Colorectal cancer ranks as the third most prevalent malignancy worldwide and the second leading cause of cancer-related mortality. For patients with locally advanced rectal cancer (LARC) classified as T3-4/N+ without distant metastasis, achieving organ preservation and functional integrity while pursuing curative treatment remains a formidable clinical challenge. This study aims to evaluate the efficacy and organ preservation rates of a novel neoadjuvant regimen comprising short-course radiotherapy followed by four cycles of CAPEOX combined with Iparomlimab and Tuvonralimab in patients with microsatellite stable (MSS) or mismatch repair proficient (pMMR) LARC. Furthermore, the project will investigate potential predictive biomarkers for complete response (CR) within this immunotherapy-based total neoadjuvant therapy (iTNT) paradigm.

DETAILED DESCRIPTION:
This study adopts a prospective, multicenter research design. It aims to evaluate the effectiveness and organ preservation rate of neoadjuvant short-course radiotherapy followed by 4 cycles of CAPEOX + Iparomlimab and Tuvonralimab in patients with MSS or pMMR LARC (AJCC eighth edition stage cT3-4 / cN+) who are initially diagnosed and can be surgically resected and randomized to the experimental group (SCRT followed by 4 cycles of CAPEOX combined with Iparomlimab and Tuvonralimab) and the control group (SCRT followed by 4 cycles of CAPEOX).

The experimental group will receive neoadjuvant short-course radiotherapy, followed by CAPEOX+Iparomlimab and Tuvonralimab for 4 cycles. The control group will receive neoadjuvant short-course radiotherapy,followed by CAPEOX for 4 cycles. During or after the completion of neoadjuvant therapy, if the patients cannot undergo radical surgical resection due to disease progression (based on RECIST v1.1) or other reasons, the treatment of this study will be terminated.

For patients who are evaluated as clinical complete remission (cCR) by imaging, colonoscopy, and pathology, the watch and wait (W&W) indications or surgical methods will be discussed by multidisciplinary team (MDT). Among them, patients with cCR or near clinical complete remission (ncCR) in efficacy evaluation will receive W&W or transanal endoscopic surgery (TES) to preserve organ function, and patients with non-cCR/ncCR will undergo total mesorectal excision (TME). After surgery, patients in the experimental group will receive CAPEOX combined with Iparomlimab and Tuvonralimab for 4 cycles, followed by sequential treatment with Iparomlimab and Tuvonralimab for up to 1 year. Patients in the control group will receive CAPEOX for 4 cycles until the planned course of treatment is completed or the disease relapses, intolerable toxicity occurs, informed consent is withdrawn, lost to follow-up or death, or other circumstances that require treatment discontinuation (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written Informed Consent Form (ICF) and be able to comply with the visits and related procedures stipulated in the protocol
2. Age between 18 and 75 years old
3. Histologically confirmed rectal adenocarcinoma
4. According to the AJCC 8th Edition staging, imaging evaluation (enhanced CT or enhanced MRI) confirms resectable locally advanced rectal cancer (AJCC 8th Edition staging cT3-4 / cN+)
5. Patients with microsatellite stability (MSS) or proficient mismatch repair (pMMR) rectal cancer
6. At least one evaluable lesion according to RECIST v1.1 criteria
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 1
8. Adequate organ and bone marrow function, defined as follows:

   * Blood count: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L; Platelet (PLT) ≥100×10^9/L; Hemoglobin (HGB) ≥10.0 g/dL.
   * Liver function: Total Bilirubin (TBIL) ≤1.5×Upper Limit of Normal (ULN); Alanine transaminase (ALT) and Aspartate transaminase (AST) ≤3×ULN. Serum albumin (ALB) ≥35 g/L.
   * Renal function: Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 ml/min (calculated using the Cockcroft-Gault formula or standard 24-hour urine collection method); Urine dipstick test shows urine protein <2+; For subjects with baseline urine dipstick test showing urine protein ≥2+, a 24-hour urine collection should be performed, and the protein content in the 24-hour urine should be <1 g.
   * Coagulation function: International Normalized Ratio (INR) ≤1.5, and Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN. Certain anticoagulant drugs (such as antiplatelet drugs, vitamin K antagonists, etc.) need to be discontinued 7~14 days before surgery and replaced with other drugs (such as low molecular weight heparin)
9. No serious concomitant diseases that threaten the subject's survival (resulting in an expected survival time of less than 5 years)
10. Female subjects of childbearing potential or male subjects with partners of childbearing potential must use effective contraception throughout the treatment period and for 6 months after the treatment period. Female subjects must have evidence of postmenopausal status or a negative urine or serum pregnancy test result for premenopausal female subjects.

Exclusion Criteria:

1. Patients with rectal cancer who have been tested for microsatellite instability as MSI-H or mismatch repair as dMMR
2. Patients who have previously received any anti-tumor treatment for the studied disease, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc. This includes previous treatment with anti-PD-1, anti-PD-L1, anti-programmed death receptor ligand 2 (PD-L2) or anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) drugs, or any other drugs acting on T cell co-stimulation or immune checkpoint pathways (such as OX40, CD137, etc.), as well as adoptive cell immunotherapy
3. Simultaneous participation in another clinical study, unless participating in an observational (non-interventional) clinical study or in the survival follow-up phase of an interventional study
4. Treatment with any investigational drug or device within 4 weeks prior to the first dose of the study drug
5. History of blood transfusion within 14 days before the screening laboratory tests, or use of Granulocyte-colony stimulating factor (G-CSF), Granulocyte-Macrophage-colony stimulating factor (GM-CSF), erythropoietin (EPO), thrombopoietin (TPO), or IL-11
6. Use of immunosuppressive drugs within 4 weeks prior to the first dose of the study drug, excluding: intranasal inhaled local steroid therapy or local steroid injections (such as intra-articular injections); systemic corticosteroid therapy not exceeding 10 mg/day of prednisone or its equivalent physiological dose; glucocorticoids as preventive medication for allergic reactions (such as pre-CT medication); use of Chinese herbal medicine or immunomodulatory drugs with anti-tumor indications (including thymosin, interferon, interleukin, etc.) within 1 week prior to the first dose of the study drug
7. Receipt of live or attenuated live vaccines within 4 weeks prior to the first dose of the study drug or expected during the study period
8. Major surgical procedures (such as craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of the study drug, anticipated need for major surgery during the study treatment period (except for radical rectal cancer surgery as specified in the protocol), or presence of unhealed wounds, ulcers, or fractures
9. Known active or suspected autoimmune disease or history of autoimmune disease within the past 2 years (subjects with eczema, vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment in the past 2 years, history of hypothyroidism requiring only thyroid hormone replacement therapy or autoimmune hypothyroidism, and type I diabetes requiring only insulin replacement therapy may be enrolled)
10. Known history of primary immunodeficiency
11. Active tuberculosis, currently receiving anti-tuberculosis treatment or having received anti-tuberculosis treatment within 1 year prior to the first dose of the study drug
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
13. Known allergy to capecitabine, oxaliplatin, anti-PD-1 monoclonal antibody, anti-CTLA-1 monoclonal antibody, anti-PD-1/CTLA-4 antibody preparation, or other monoclonal antibody components
14. Ascites and pleural effusion requiring clinical intervention in the short term, symptomatic or requiring drainage of pericardial effusion
15. Human immunodeficiency virus (HIV) infection (HIV antibody positive)
16. Acute or chronic active hepatitis B (defined as HBsAg or only HBcAb positive and HBV DNA ≥2000 IU/mL or ≥1×10^4 copies/mL), acute or chronic active hepatitis C (defined as HCV antibody positive and HCV-RNA level above the lower limit of detection)
17. HBV DNA ≥2000 IU/mL or ≥1×10^4 copies/mL), acute or chronic active hepatitis C (defined as HCV antibody positive and HCV-RNA level above the lower limit of detection)
18. Active syphilis infection requiring treatment
19. Severe infection occurring within 4 weeks prior to the first dose of the study drug or during the active phase or poorly controlled, including but not limited to hospitalization for infection, bacteremia, or complications of severe pneumonia, therapeutic oral or intravenous antibiotics within two weeks prior to the first dose
20. Symptomatic congestive heart failure (New York Heart Association class II~IV) or left ventricular ejection fraction (LVEF) <50% on echocardiography; symptomatic or poorly controlled arrhythmia; history of congenital long QT syndrome or corrected QTc >500 ms at screening (calculated using Fridericia's method)
21. Uncontrolled arterial hypertension despite standard treatment (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg), history of hypertensive crisis or hypertensive encephalopathy
22. Severe bleeding tendency or coagulation dysfunction, or undergoing thrombolytic therapy
23. Any arterial thromboembolic event within 6 months prior to the first dose of the study drug, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack
24. Esophageal or gastric varices requiring immediate intervention (e.g., ligation or sclerotherapy) or considered at high risk of bleeding by the investigator or after consultation with a gastroenterologist or hepatologist, evidence of portal hypertension (including splenomegaly on imaging) or history of variceal bleeding, subjects must undergo endoscopic evaluation within 3 months prior to enrollment
25. History of gastrointestinal perforation and/or fistula within 6 months prior to the first dose of the study drug
26. Any life-threatening bleeding event within 3 months prior to the first dose of the study drug, or grade 3 or 4 gastrointestinal/variceal bleeding event requiring transfusion, endoscopy, or surgical treatment
27. History of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolic event within 3 months prior to the first dose of the study drug (implantable venous port or catheter-related thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism)
28. Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or cancer-related reactions that may lead to higher medical risks and/or uncertainty in survival evaluation
29. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B >7 points or more severe cirrhosis
30. Intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition) and not relieved by the screening period; subjects at risk of intestinal perforation (including but not limited to acute diverticulitis, abdominal abscess, history of abdominal cancer); history of extensive intestinal resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea
31. Interstitial lung disease requiring treatment; history and current presence of pulmonary fibrosis, pneumoconiosis, drug-related pneumonia, organic pneumonia (such as bronchiolitis obliterans), severe pulmonary impairment, etc.
32. Significant malnutrition (weight loss of 5% within 1 month or 15% within 3 months prior to signing the informed consent, or reduction in food intake by 1/2 or more within 1 week), or patients requiring intravenous nutritional support. However, malnutrition corrected more than 4 weeks prior to the first dose of the study drug is excluded
33. History of other primary malignancies, except: malignancies that have been cured, with no known active disease for ≥2 years prior to the first dose of the study drug and with a very low risk of recurrence
34. Adequately treated non-melanoma skin cancer or malignant lentigo with no evidence of disease recurrence
35. Adequately treated carcinoma in situ with no evidence of disease recurrence
36. Other acute or chronic diseases that may result in: increased risk related to study participation or study drug administration, or interference with the interpretation of study results, and in the investigator's judgment, render the subject ineligible for participation in this study
37. Neurological, psychiatric disorders, or social conditions that: affect compliance with study requirements, significantly increase the risk of adverse events, or affect the subject's ability to provide written informed consent, such as history of schizophrenia, drug abuse, etc.
38. Alcohol, drug, or substance use that may hinder drug administration or affect toxicity analysis
39. Pregnant or breastfeeding female subjects
40. Other situations deemed unsuitable for enrollment by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response | From date of randomization until the date of treatment of surgery, assessed up to 5 months
Clinical Complete Response | From date of randomization until the date of discussion of multidisciplinary team, assessed up to 5 months
Pathologic Complete Response | From date of randomization until the date of treatment of surgery, assessed up to 5 months

SECONDARY OUTCOMES:
Organ Preservation Rate | From date of randomization until the date of treatment of additional surgery, assessed up to 100 months
Major Pathologic Response | From date of randomization until the date of treatment of surgery, assessed up to 5 months
Overall Surviral | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
Desease Free Survival | From date of randomization until the date of first documented progression, whichever came first, assessed up to 100 months
Anal Sphincter Preservation Rate | From date of randomization until the date of treatment of surgery, assessed up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Guosheng Wu, MD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No